CLINICAL TRIAL: NCT05983614
Title: Investigation of the Effects of Pain, Proprioception and Electrodiagnostic Findings on Activity and Participation in Patients With Idiopathic Carpal Tunnel Syndrome
Brief Title: Effects of Body Structures and Function on Actıvıty and Partıcıpatıon in Patıents wıth Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Head of Occupational Therapy Deparment, Kutahya Health Sciences University
Other Study IDs: 2022/16-2
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Pain; Proprioception; Sensation; EMG; ICF
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to determine pain, sensation and electrodiagnostic findings in CTS; to examine its effects on activity and participation.

DETAILED DESCRIPTION:
50 patients aged 20-55 years diagnosed with mild and moderate carpal tunnel syndrome according to AANEM will be included. VAS, LANSS, Boston Carpal Tunnel Questionnaire (Symptom Severity Scale - Functional Status Scale), Q-DASH, hand grip sensitivity measurement, hand pressure sensitivity measurement will be applied to the participants. In order to examine the relationship between body structure and functions (Pain, Sensation, EMG findings) and activity and participation with the AMOS program, the maximum likelihood method will be selected and a structural equation model (SEM) will be established.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mild-moderate CTS
* Being between the ages of 20-55
* Volunteering to participate in the study

Exclusion Criteria:

* Being diagnosed with severe CTS
* Have systemic inflammatory disease
* Having a disease that can cause polyneuropathy, such as diabetes mellitus
* Being receiving psychotherapy
* Illiteracy
* Have a hearing problem
* Have cognitive impairment
* Having a pacemaker

Ages: 25 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Patients who applied to the Physical Therapy Department of Kutahya Health Sciences University Hospital and were diagnosed with mild and moderate CTS according to the American Association of Neuromuscular and Electrodiagnostic Medicine (AANEM) will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Leeds Assessment Neuropathic Symptoms and Signs (LANSS) | 7 minutes
  Leeds Assessment Neuropathic Symptoms and Signs (LANSS) scale is a clinical-based tool for identifying pain and patients with predominant neuropathic mechanisms.
Boston Carpal Tunnel Questionnaire | 12 minutes
  It is a questionnaire used to evaluate symptom severity and functional status in individuals with carpal tunnel syndrome.
Q-DASH | 10 minutes
  Q-DASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.

SECONDARY OUTCOMES:
Proprioception Assessment | 7 minutes
  Hand grip sensitivity will be measured with a dynamometer and hand pressure sensitivity will be measured with a Stabilizer Pressure Biofeedback (SBP) instrument.
Visual Analog Scale | 2 minutes
  Evaluates the severity of pain, scoring between 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Afsar, Phd, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)